CLINICAL TRIAL: NCT02460120
Title: Evaluation of the Archimedes™ System for Transparenchymal Nodule Access
Acronym: EAST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Updates to device
Sponsor: Broncus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Protocol 43
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Navigation and tissue sampling (Experimental): Guided bronchoscopic navigation and lung tissue sampling using the Archimedes System
  Interventions: Device: Archimedes System

INTERVENTIONS:
Device: Archimedes System — The Archimedes System is an image-guided navigation system used to access tissue samples in the lungs

SUMMARY:
The Archimedes System is an image-guided navigation system used to access tissue samples in the lungs. This study is being conducted to confirm the performance of the Archimedes System in patients who are scheduled for standard bronchoscopy to diagnose highly suspicious lung cancer or metastatic disease. Navigation to and sampling of the patient's lung cancer tumor is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-75 years at screening
2. Highly suspicious SPN, defined as distinct nodule with a diameter of ≥8mm in its largest dimension
3. No known endobronchial tumor
4. Tumor located anywhere in parenchymal tissue >1 cm from pleura and accessible bronchoscopically through a POE.
5. Willing to participate in all aspects of study protocol for duration of study
6. Able to understand study requirements
7. Signs study-related informed consent document

Exclusion Criteria:

1. Any contraindication to bronchoscopy, for example:

   * Untreatable life-threatening arrhythmias
   * Inability to adequately oxygenate the patient during the procedure
   * Acute respiratory failure with hypercapnia (unless the patient is intubated and ventilated)
   * Recent myocardial infarction
   * Previously diagnosed high-grade tracheal obstruction
   * Uncorrectable coagulopathy
2. Known coagulopathy
3. Platelet dysfunction or platelet count < 100 x 103 cells/mm3
4. History of major bleeding with bronchoscopy
5. Suspected pulmonary hypertension: additional testing required, such as echocardiogram
6. Moderate-to-severe pulmonary fibrosis
7. Severe emphysema or COPD: additional testing and PI consent is required
8. Bullae >5 cm located in vicinity of target SPN
9. Any other severe or life-threatening comorbidity that could increase the risk of bronchoscopic biopsy or ATV tunneling, for example:

   * ASA class > 3
   * > stage 3 heart failure
   * severe cachexia
   * severe respiratory insufficiency or hypoxia
10. Ongoing systemic infection
11. Contraindication to general anesthesia
12. Inability to stop anticoagulants (e.g., heparin, Warfarin) or antiplatelet agents (e.g. aspirin, clopidogrel) prior to procedure
13. Participation in any other study in last 30 days
14. Prior thoracic surgery on the same side of the lung as the SPN.
15. Breastfeeding women or females of childbearing potential with a positive pregnancy test prior to the procedure or the intent to become pregnant during the study.
16. Life expectancy of less than one year.
17. Scheduled for lung surgery within 72hrs post-scheduled diagnostic bronchoscopy
18. Pregnancy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of biopsies yielding tissue sufficient for diagnosis | Up to 1 year
  The the number of nodules with at least one biopsy sufficient for a definitive tissue diagnosis divided by the number of nodules sampled by the Archimedes System.

SECONDARY OUTCOMES:
Procedure planning time | Up to 1 year
  The time from selecting the patient CT until the tunnel path has been selected, reviewed and exported.
Nodule access time | Up to 1 year
  The time from the start of navigation until the sheath has been placed at the first biopsy target.
Fluoroscopy time | Up to 1 year
  The total fluoroscopy time from the start of fused-fluoroscopic navigational guidance to the time the devices are removed from the point of entry.
Patient registration time | Up to 1 year
  The total time it takes to correlate the patient's position via fluoroscopy with the navigational guidance system.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Nader, D.O., Principal Investigator — Cancer Treatment Centers of America at Southwestern Regional Medical Center
Locations (1):
- Cancer Treatment Centers of America at Southwestern Regional Medical Center, Tulsa, Oklahoma, United States